CLINICAL TRIAL: NCT05653349
Title: A Phase III, Randomized, Double-blind Study of Ianalumab (VAY736) Versus Placebo in Addition to First-line Corticosteroids in Primary Immune Thrombocytopenia (VAYHIT1)
Brief Title: Study of Ianalumab Versus Placebo in Addition to First-line Corticosteroids in Primary Immune Thrombocytopenia (ITP)
Acronym: VAYHIT1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736I12301
Record Dates: First submitted 2022-11-23; First posted 2022-12-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: Primary immune thrombocytopenia (ITP); ianalumab; VAY736; B-cell depletion; B-cell Activating Factor Receptor (BAFF-R) blockade
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — ianalumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ianalumab Lower dose (Experimental): Lower dose of ianalumab administered intravenously with corticosteroids oral or parental (if clinically justified)
  Interventions: Biological: Ianalumab; Drug: Corticosteroids
- Ianalumab Higher dose (Experimental): Higher dose of ianalumab administered intravenously with corticosteroids oral or parental (if clinically justified)
  Interventions: Biological: Ianalumab; Drug: Corticosteroids
- Placebo (Placebo Comparator): Placebo administered intravenously with corticosteroids oral or parental (if clinically justified)
  Interventions: Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Biological: Ianalumab — Intravenous infusion, prepared from concentrate solution
  Other Names: VAY736
  Arms: Ianalumab Higher dose; Ianalumab Lower dose
Drug: Placebo — Intravenous infusion, prepared from matching placebo
  Arms: Placebo
Drug: Corticosteroids — Oral or parental (if clinically justified)

SUMMARY:
The purpose of this study is to evaluate the effect of two different doses of ianalumab versus placebo in addition to first-line corticosteroids in maintaining platelet count ≥30 G/L in adult participants with primary ITP.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind Phase 3 study to assess the efficacy and safety of two different doses of ianalumab compared to placebo in adults with primary ITP (platelets count <30 G/L) who require first-line standard-of-care corticosteroids.

After completion of the screening period, the participants will enter the randomized treatment period (ianalumab/placebo with standard of care corticosteroids).

After the treatment period, all participants will enter the follow-up period to be monitored for efficacy and safety or safety only depending on how they respond to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation in the study.
* Male or female participants aged 18 years and older on the day of signing informed consent
* Primary ITP diagnosed within 3 months before initiating first-line ITP therapy (corticosteroids, IVIG)
* Platelet count below 30 G/L before starting any first-line ITP therapy (corticosteroids, IVIG)
* Response (platelet count >=50 G/L) to corticosteroids (+/- IVIG) at any time prior to randomization. Note: Platelet count measured within 7 days of platelet transfusion will not be considered as response.

Key Exclusion Criteria:

* Evans syndrome or any other cytopenia (patients with low grade anemia related to bleeding or iron deficiency are eligible)
* Current life-threatening bleeding
* Previous ITP treatment, including splenectomy, except for corticosteroids and/or IVIG initiated as first-line therapy for up to 28 days before randomization and rescue corticosteroids and/or IVIG given prior to confirmed diagnosis of primary ITP .
* Prior use of B-cell depleting therapy (e.g., rituximab).
* Absolute neutrophil count below 1.0 G/L at randomization
* Participants with concurrent coagulation disorders and/or receiving anti-platelet or anticoagulant medication with an exemption of low dose of acetylsalicylic acid

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to treatment failure (TTF) | Randomization to end of study (up to 39 months after randomization of last patient)
  Time from randomization until platelet count below 30 G/L, need for a rescue treatment or start of a second-line therapy or death.

SECONDARY OUTCOMES:
Complete Response (CR) rate in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Complete Response (CR) rate at each timepoint defined as the proportion of participants with any platelet count of at least 100 G/L in the absence of rescue treatment or new ITP treatment.
Response (R) rate in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Response (R) rate at each timepoint defined as the proportion of participants with any platelet count of at least 50 G/L in the absence of rescue treatment or new ITP treatment.
Time to complete response in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Time from randomization to date of first complete response.
Duration of response in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Time from achievement of complete response to loss of complete response
Stable response at 6 months | At 6 months
  Percentage of participants with at least 2 platelet count collected at month 6 (between study dates 107 and 183) and at least 66% of platelet counts qualified as a response
Stable response at 1 year | At 1 year
  Percentage of participants with at least 2 platelet counts collected at year 1 (between study days 296 and 379) and at least 66% of platelet counts qualified as a response
Percentage of participants with bleeding events overall and by World Health Organization (WHO) bleeding scale severity | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the incidence and severity of bleeding in each treatment arm
Number of participants with bleeding events overall and by World Health Organization (WHO) bleeding scale severity | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the number and severity of bleeding in each treatment arm
Number of participants receiving rescue treatment (cummulative dose/duration of steroids exposure) | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the number of participants receiving rescue treatment.
Percentage of participants receiving rescue treatment (cummulative dose/duration of steroids exposure) | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the need of rescue treatment in each treatment group by percentage.
Cumulative dose/duration of steroids exposure | From screening to end of study (up to 39 months after randomization of last patient)
  Duration of exposure to corticosteroids calculated from randomization (first dose) to end of study or last last contact date (if the participant is lost to follow-up).
Change from baseline on T scores of the PROMIS SF v1.0 Fatigue 13a | From screening (baseline) till end of study (up to 39 months after randomization of last patient)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Fatigue 13a includes 13 items that assess fatigue
Change from baseline in ITP-PAQ domain scores | From screening (baseline) till end of study (up to 39 months after randomization of last patient)
  The ITP-PAQ is a 44 item scale for measuring HRQoL in adults with ITP across ten scales: Symptoms, Bother-Physical Health, Fatigue/Sleep, Activity, Fear, Psychological Health, Work, Social Activity, Women's Reproductive Health, and Overall QoL. Each item is rated on a Likert type scale
Change from baseline in frequency of CD19+ B cell counts | Randomization to end of study (up to 39 months after randomization of last patient)
  Post baseline frequency (%within the CD45) of CD19+ B cell counts compare to baseline.
Change from baseline in absolute number of CD19+ B cell counts | Randomization to end of study (up to 39 months after randomization of last patient)
  Post baseline absolute number of CD19+ B cell counts compare with baseline
Time to first occurrence of B-cell recovery | Randomization to end of study (up to 39 months after randomized of last patient)
  B-cell recovery, defined as ≥80% of baseline or ≥50 cells/μL
Change from baseline in inmmunoglobulins | Randomization to end of study (up to 39 months after last randomized patients)
  Change from baseline in immunoglobulin levels
PK parameters: AUClast | After first dose (pre-dose, 2, 168, 336 and 504 hours post dose) and after last dose (pre-dose, 2, 336, 672, 1344, 2016, 3360 hours post dose)
  AUClast: area under the curve from time zero till the last measurable concentration sampling time (tlast)
PK parameter: AUCtau | After first dose (pre-dose, 2, 168, 336 and 504 hours post dose) and after last dose (pre-dose, 2, 336, 672, 1344, 2016, 3360 hours post dose)
  Area under the curve calculated to the end of a dosing interval (tau)
PK parameters: Cmax | After first dose (pre-dose, 2, 168, 336 and 504 hours post dose) and after last dose (pre-dose, 2, 336, 672, 1344, 2016, 3360 hours post dose)
  Maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration
PK parameters: Tmax | After first dose (pre-dose, 2, 168, 336 and 504 hours post dose) and after last dose (pre-dose, 2, 336, 672, 1344, 2016, 3360 hours post dose)
  Time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration
PK parameters: Accumulation ratio Racc | After last dose (pre-dose, 2, 336, 672, 1344, 2016, 3360 hours post dose)
  Accumulation ratio calculated using AUC values obtained between the last and first dose
Incidence of anti-ianalumab antibodies in serum (ADA assay) over time | Up to Week 33
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants assess the immunogenicity of ianalumab
Titer of anti-ianalumab antibodies in serum (ADA assay) over time | Up to Week 33
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants assess the immunogenicity of ianalumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (114):
- United States (21):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Community Cancer Institute, Clovis, California
  - Compassionate Care Res Group Inc, Fountain Valley, California
  - University of Colorado Anschutz, Aurora, Colorado
  - DH Cancer Research Center LLC, Margate, Florida
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Oncology Care Associates, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Clinical Research Alliance, Lake Success, New York
  - Hematology Oncology Association of Rockland, Nyack, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - STAT Research Inc, Dayton, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Córdoba
- Australia (4):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Salzburg
- Belgium (4):
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Leuven
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- China (16):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Luoyang, Henan
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Xi'an, Shaanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Bengbu
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Tianjin
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- France (4):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Chambéry
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Rennes
- Germany (6):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Giessen
- Hong Kong (2):
  - Novartis Investigative Site, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- India (4):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Rishikesh, Uttarakhand
  - Novartis Investigative Site, Kolkata, West Bengal
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Vicenza, VI
- Japan (9):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Shibukawa, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Osaka
- Malaysia (4):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, George Town
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Selangor
- Mexico (4):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Mexico City, Mexico CP
  - Novartis Investigative Site, Morelia, Michoacán
  - Novartis Investigative Site, Monterrey, Nuevo León
- Novartis Investigative Site, Grålum, Norway
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Singapore, Singapore
- Spain (5):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Aydin, Efeler
  - Novartis Investigative Site, Istanbul, Fatih
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com